CLINICAL TRIAL: NCT03566589
Title: Effects of Lactobacillus Plantarum PS128 on the Parkinsonian Symptoms in Parkinson's Disease: a Pilot Study
Brief Title: Effects of PS128 on Parkinsonian Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Professor Lu Neurological Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PS128-01
Record Dates: First submitted 2018-06-12; First posted 2018-06-25 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PS128 (Experimental): daily ingestion of Lactobacillus plantarum PS128 capsules
  Interventions: Dietary Supplement: Lactobacillus plantarum PS128

INTERVENTIONS:
Dietary Supplement: Lactobacillus plantarum PS128 — daily ingestion of 60 billion colony forming unit (CFU) of Lactobacillus plantarum PS128 (30 billion CFU/capsule)
  Other Names: PS128

SUMMARY:
The purpose of this study is to examine the short term effects (12 Weeks) of Lactobacillus plantarum PS128 (PS128) on Parkinson's disease (PD) symptoms.

DETAILED DESCRIPTION:
This study is designed to examine the extent to which L. plantarum PS128 can improve symptoms in PD patients. L. plantarum PS128 is a psychobiotic that regulates the level of dopamine in specific brain regions. Patients with PD will receive PS128 treatment for 12 weeks. Symptoms of PD will be clinically evaluated before and after the treatment, and the results will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Between ages of 40-80 years old
* Diagnosed as a patient with Parkinson's disease of modified Hoehn and Yahr Stage between 1 and 2.5 as rated during an "on" period

Exclusion Criteria:

* Patients on antibiotics within the preceding one month
* Patients using of other probiotic products (sachet, capsule or tablet) within the preceding two weeks
* Have current or history of inflammatory bowel disease
* Have history of cancer
* Have undergone surgery of liver, bladder, or gastrointestinal tract
* Known allergy to probiotics
* Patients with comorbid dementia (Mini-Mental State Examination score ≤ 26) or major depression (The Beck Depression Inventory-II score ≥ 29)
* Have received deep brain stimulation
* Patients receiving artificial enteral or intravenous nutrition

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-07-02 (Actual); Primary Completion 2018-11-09 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Change in Unified Parkinson's Disease Rating Scale (UPDRS) Score From Baseline to Change in Unified Parkinson's Disease Rating Scale (UPDRS) (Part III) Motor Score From Baseline to Week 12 Assessed On Medication | Baseline to Week 12
  The UPDRS scores is a rating tool used to gauge the course of Parkinson's disease in patients. The minimum total score possible is 0 and the maximum total score possible is 199. Higher values represent a worse outcome.

SECONDARY OUTCOMES:
Change in Nonmotor Symptoms: 30-item Screening Questionnaire (NMS-Quest) Score From Baseline to Week 12 Assessed On Medication | to Week 12 Assessed On Medication
  NMS-Quest is a 30-item Screening tool for non-motor symptoms of Parkinson's disease. The minimum total score possible is 0 and the maximum total score possible is 30. Higher values represent a worse outcome.
Change in Patient Global Impression of Change (PGIC) Score From Baseline to Week 12 Assessed On Medication | to Week 12 Assessed On Medication
  The PGIC consists of one item taken from the clinical global impression and adapted to the patient. The minimum total score possible is 1 and the maximum total score possible is 7. Higher values represent a worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Professor Lu Neurological Clinic, Taoyuan, Guishan Dist., Taiwan

IPD SHARING:
Plan to Share IPD: No